CLINICAL TRIAL: NCT03908866
Title: Peripherally Inserted Versus Centrally Inserted Central Venous Catheters in the Neurosurgical Intensive Care Unit. Comparative of Cost-Effectiveness and Safety
Brief Title: Peripherally Inserted Versus Centrally Inserted Central Venous Catheters in the Neurosurgical Intensive Care Unit
Acronym: PICINI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: XJTU1AF2019LSK-2019-032
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Thromboses, Venous; Infection; Economic Problems
MeSH Terms: conditions — Venous Thrombosis; Infections | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICC(Peripherally inserted central catheter) (Experimental): Patients randomly assigned to receive a peripherally inserted central catheter(PICC).
  Interventions: Other: PICC(Peripherally inserted central catheter)
- CVC(Central venous catheter ) (Active Comparator): Patients randomly assigned to receive a centrally inserted central venous catheter(CVC).
  Interventions: Other: CVC(Central venous catheter )

INTERVENTIONS:
Other: PICC(Peripherally inserted central catheter) — The peripherally inserted central catheter with different sizes (French scale). Trained vascular access nurses will perform the insertion of the PICC, guided by ultrasound at bedside using the Seldinger technique. A suitable sterile field will be established.
  Arms: PICC(Peripherally inserted central catheter)
Other: CVC(Central venous catheter ) — The central venous catheter with different sizes (French scale). Trained doctors will perform the insertion of the CVC, using the Seldinger technique. A suitable sterile field will be established.
  Arms: CVC(Central venous catheter )

SUMMARY:
This study aim to compare the cost-effectiveness and safety between centrally and peripherally inserted central venous catheters in neurosurgical intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the neurosurgical intensive care unit , who require central access for the treatment of their illness.

Exclusion Criteria:

* Insertion of the central catheter in emergency situations;
* Anatomical abnormalities of upper extremity affecting PICC placement;
* Current or recent (within 1 month) diagnosis of bacteremia
* Current or recent (within 1 year with confirmed resolution by imaging) deep venous thrombosis;
* Presence of skin changes in the area of the puncture, such as thrombophlebitis, dermatitis, cellulitis, burn among others;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
thrombotic complications | up to 30 days or be discharged from hospital
  radiographically-confirmed upper-extremity deep vein thrombosis
mechanical complications | up to 30 days or be discharged from hospital
  pneumothorax or hematoma caused by puncture
infectious complications | up to 30 days or be discharged from hospital
  catheter related bloodstream infection

SECONDARY OUTCOMES:
catheter replacement | up to 30 days or be discharged from hospital
  obstruction or accidental removal
cost effectiveness | up to 30 days or be discharged from hospital
  The cost of catheter implantation and replacement, as well as the cost of treatment due to catheter-related complications and the resulting financial loss to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Liu, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China